CLINICAL TRIAL: NCT00401557
Title: Intervenable Host - Leishmania (Viannia) Interactions - Project 3: Immune and Inflammatory Responses in L. (Viannia) Infection - Aim 3: Mechanisms Relating to the Distinct in Vitro Susceptibility of Human Macrophages to L. Viannia Infection
Brief Title: Mechanisms Relating to the Distinct in Vitro Susceptibility of Human Macrophages to L. Viannia Infection
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Dr. Diane McMahon-Pratt, Yale University
Other Study IDs: 0608001740; U19AI065866 (NIH)
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2011-08

CONDITIONS: Leishmaniasis
Keywords: Leishmaniasis, Leishmania (Viannia), Colombia
MeSH Terms: conditions — Leishmaniasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine how the body defends itself against Leishmania (Viannia), a parasite that can cause a skin infection and skin sores. Certain cells in the immune system act more aggressively against Leishmania in people with mild Leishmania symptoms than in those who have long-term or recurring symptoms of the disease. Participants in the study will include people who currently have Leishmania infection, people who have had the infection in the past, and people who have never been exposed to the parasite. This study will enroll 220 adults, ages 18 to 70 years, at 3 sites in Colombia. Blood samples will be collected from volunteers at least once during the study. Participants will also undergo HIV testing. Volunteers will participate in up to 2 study visits, scheduled 2-3 weeks apart.

DETAILED DESCRIPTION:
This is a cross-sectional study that aims to determine the mechanisms that lead to the distinct in vitro susceptibility of human macrophages to L. Viannia infection, and their relationship to clinical phenotype. It is the third part of a study which includes DMID protocols 06-0009 and 06-0010. The general objective of the study is to determine the mechanisms that lead to the distinct in vitro susceptibility of human macrophages to L. Viannia infection, and their relationship to clinical phenotype. (Understanding the immune mechanisms underlying disease should provide insight for the development of new methods for treatment and intervention.) The specific objectives of the study are: to determine the association of the Toll response profile of monocytes and macrophages with the in vitro susceptibility phenotype, and analyze Toll receptor response in relation with both in vitro and clinical phenotype in participants presenting asymptomatic, chronic and recurrent disease and in healthy donors (controls)(Toll receptors); to determine gene expression response of susceptible and resistant macrophages to exposure and infection by L. panamensis, in order to identify genes and gene products that determine the course of infection in the host cell and that are linked to clinical response; to define the interaction of cytokines and Leishmania infection in promoting the latent persistence of infection or activation of growth, and to explore the role of apoptosis in elimination or propagation of infection (Apoptosis); and to determine the functional phenotypic characteristics of susceptible and resistant macrophages from healthy donors and clinically disparate individuals by flow cytometric analyses (Functional Phenotype of mononuclear phagocytes). Participants of the four specific objectives will be asked to provide relevant demographic, clinical and epidemiologic information and blood samples. Monocytes and macrophages differentiated from peripheral blood samples will be analyzed by different methodologies (flow cytometry, Real time PCR, ELISA and microarray analysis), and the results compared across the groups in order to determine if the macrophage response to infection is a determinant of recurrent and/or chronic disease development. Participants will be enrolled at three sites in Colombia: CIDEIM, Cali; CIDEIM, San Andrés Hospital, Tumaco; and San Juan Bautista Hospital, Chaparral. Patients (males and females) aged between 18-70 years with historic chronic or recurrent cutaneous leishmaniasis diagnosed at any of these three study sites will be invited to participate in the study. Asymptomatic and healthy donors (controls) will also be enrolled. A maximum of 220 participants will be enrolled. For historic (chronic and recurrent) and asymptomatic participants, a single study visit is planned. For healthy donors, 2 study visits are planned. The second visit will be programmed 2-3 weeks after the first visit. Study outcome measures will be levels of transcription of cytokines (e.g. TNF-alpha, IL-10, IL-12) and nuclear transcription factors normalized to the number of macrophages; percentage of non-infected and infected macrophages/monocytes expressing specific cytokine receptors and Toll like receptors; density of receptor expression; percentage of apoptotic cells; number and change in number of parasites in apoptotic and non-apoptotic cells; nitric oxide level; cytokine production as concentration of supernatants of macrophage cultures (e.g. TNF-alpha, IL-10, and IL-12); intracellular cytokine production, intracellular nitric oxide level; percentage of infected macrophages/monocytes and number of intracellular parasites over time to assess survival and replication; and percentage of non-infected and infected macrophages/monocytes expressing specific activation and differentiation markers and the intensity of marker expression.

ELIGIBILITY:
Inclusion Criteria:

For specific objectives 1, 3 and 4:

Historical cases of chronic disease:

* Age between 18-70 years
* Historic parasitologically confirmed, skin test positive cutaneous leishmaniasis (CL) patients who presented chronic CL lesions of > 6 months duration at the time of diagnosis
* No active lesions
* Voluntary participation in the study
* Written and signed Informed consent for HIV testing and participation in the study

Historical cases of recurrent disease:

* Age between 18-70 years
* Historic CL patients who have developed new parasitologically confirmed lesions after resolution of prior disease
* No active lesions
* Voluntary participation in the study
* Written and signed Informed consent for HIV testing and participation in the study

Asymptomatic infection:

* Age between 18-70 years
* Resident of endemic area
* No history or evidence of active or prior dermal leishmaniasis
* Voluntary participation
* Written and signed Informed consent for HIV testing and participation in the study

Healthy donors:

* Age between 18-70 years
* No history or evidence of exposure to transmission of leishmaniasis
* Voluntary participation
* Written and signed Informed consent for HIV testing and participation in the study

For specific objective 2:

Historical cases of chronic disease:

* Age between 18-70 years
* Historic parasitologically confirmed, skin test positive CL patients who presented chronic CL lesions of > 6 months duration at the time of diagnosis
* No active lesions
* Voluntary participation in the study
* Written and signed Informed consent for HIV testing and participation in the study

Historical cases of recurrent disease:

* Age between 18-70 years
* Historic CL patients who have developed new parasitologically confirmed lesions after resolution of prior disease
* No active lesions
* Voluntary participation in the study
* Written and signed Informed consent for HIV testing and participation in the study

Asymptomatic infection:

* Age between 18-70 years
* Resident of endemic area
* No history or evidence of active or prior dermal leishmaniasis
* Voluntary participation
* Written and signed Informed consent for HIV testing and participation in the study

Healthy donors:

* Age between 18-70 years
* No history or evidence of exposure to transmission of leishmaniasis
* Voluntary participation
* Written and signed Informed consent for HIV testing and participation in the study

Exclusion Criteria:

Exclusion criteria for all groups (for specific objectives 1, 3 and 4):

* Immunosuppressive disease
* Pharmacotherapy with drugs that are immunosuppressive
* Pregnancy
* Breastfeeding
* Unwillingness to participate

Exclusion criteria for all groups (for specific objective 2):

* Weight below 50kg
* Immunosuppressive disease (HIV)
* Treatment with drugs that are immunosuppressive
* Pregnancy
* Breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Historical cases of chronic disease:
  * Age between 18-70 years
  * Historic parasitologically confirmed, skin test positive cutaneous leishmaniasis (CL) patients who presented chronic CL lesions of > 6 months duration at the time of diagnosis
  * No active lesions
  Historical cases of recurrent disease:
  * Age between 18-70 years
  * Historic CL patients who have developed new parasitologically confirmed lesions after resolution of prior disease
  * No active lesions
  Asymptomatic infection:
  * Age between 18-70 years
  * Resident of endemic area
  * No history or evidence of active or prior dermal leishmaniasis
  Healthy donors:
  * Age between 18-70 years
  * No history or evidence of exposure to transmission of leishmaniasis
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2006-12; Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Saravia, Ph.D., Principal Investigator — Centro Internacional de Entrenamiento e Investigaciones Médicas
Locations (1):
- Centro Internacional de Entrenamiento e Investigaciones Medicas, CIDEIM, Cali, Colombia